CLINICAL TRIAL: NCT00730366
Title: New Approaches to Improve Coverage and Compliance of Antimalarial Treatment for Pregnant Women in Rural Africa.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University of Ouagadougou, Burkina Faso (Other); National Laboratory of Public Health,Burkina Faso (Unknown); Liverpool School of Tropical Medicine (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Prof. Umberto D'Alessandro, Institute of Tropical Medicine, Antwerp, Belgium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DELIMAL
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Malaria in Pregnancy
Keywords: Malaria; Pregnancy; Intermittent Preventive Treatment
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Experimental: IPTp-SP + promotion: Active Comparator
  Interventions: Drug: sulfadoxine-pyrimethamine
- 2 (Experimental): IPTp-SP alone (without promotion)
  Interventions: Drug: sulfadoxine-pyrimethamine
- 3 (Active Comparator): Weekly CQ prophylaxis
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine — Sulfadoxine-pyrimethamine given as intermittent therapy, at the dosage of 1500/75 mg per administration (3 tablets), Twice during pregnancy
  Other Names: IPTp-SP, SP, Fansidar
  Arms: 1; 2
Drug: Chloroquine — Chloroquine tablets 100 mg. First administration of 1500 mg given over three days, followed by weekly doses of 300 mg/week
  Other Names: CQ, Nivaquine
  Arms: 3

SUMMARY:
Malaria in pregnancy contributes substantially to maternal anaemia and low birth weight: effective malaria control in pregnancy could avoid about 10,000 maternal and up to 200,000 infant deaths every year. Intermittent preventive treatment with the drug sulfadoxine-pyrimethamine (IPTp-SP), administered at least twice during routine antenatal clinics, is recommended by the World Health Organization for areas of moderate to high malaria transmission, including Sub-Saharan Africa.

Studies carried out in Kenya and Malawi before 2004 had showed that two doses of IPTp-SP significantly reduce maternal anaemia, placental malaria parasitaemia and low birth weight. However, in countries where this strategy had been introduced as part of national policy, the coverage of the target population has varied widely, with estimates of 33-93% for uptake of one dose and 24-68% for two doses, and no country had reached the goal of 80% of pregnant women receiving at least 2 doses of IPTp. New approaches designed to improve IPTp coverage were therefore urgently needed.

This study was therefore set up in 2002, in order to evaluate the additional effect of a targeted promotional campaign on antenatal clinics utilization and on coverage and uptake of Intermittent preventive treatment with sulfadoxine-pyrimethamine in a rural health district in Burkina Faso; and to investigate the effectiveness of intermittent preventive treatment with the sulfadoxine-pyrimethamine compared with weekly chloroquine, in order to provide additional evidence to the Burkinabé Ministry of Health for an impending policy change.

DETAILED DESCRIPTION:
Each year, about 50 million women living in malaria endemic regions become pregnant, more than half in sub-Saharan Africa. In areas of relatively stable transmission, where acquired immunity to Plasmodium falciparum limits infection and prevents severe disease in adults, women in their first and second pregnancy are the most vulnerable subjects, due to a higher risk of severe anaemia and a low birth weight (LBW) outcome, a leading cause of child mortality and poor growth and development.

Malaria in pregnancy and its adverse consequences can be prevented with suppressive antimalarial treatment or chemoprophylaxis. Weekly chloroquine (CQ) had been the basis for prevention for many years, but its application became limited over time, partly because of difficulties in coverage and compliance throughout pregnancy and partly because of increased parasite resistance to CQ in endemic areas. A new strategy for prevention based on insecticide-treated bed nets (ITNs) and use of intermittent preventive treatment in pregnancy (IPTp) was thus formulated, with IPTp being based on the administration of treatment doses of sulfadoxine-pyrimethamine (1500/75 mg; SP) to all pregnant women at pre-defined intervals and regardless of malaria infection. WHO elaborated new recommendations, based on the administration of SP two or three times at scheduled antenatal visits at least one month apart from the second trimester onwards. Evidence of the efficacy of IPTp with SP for preventing malaria infection and improving birth weight was reported from East Africa and West Africa.

However, the IPTp strategy assumes that most pregnant women attend antenatal clinics (ANC) at least twice during their pregnancy and at a time when SP can be administered under direct observation. Unfortunately, it appeared soon that late attendance to ANC and weak health services limit the effectiveness of this strategy; coverage with two or more SP doses varied widely (24-68%) and was well behind the goal of 80% proposed by the Roll Back Malaria Partnership. New approaches to increase IPTp coverage were urgently needed.

This study, conceived in 2002 and carried out between 2004 and 2006, had therefore two different components: on one side, it investigated whether promoting regular and early antenatal attendance of pregnant women through community based health education would increase coverage and uptake of IPTp; on the other side, it investigated the effectiveness of IPTp-SP compared with weekly CQ, in order to provide additional evidence to the Burkinabé Ministry of Health for an impending policy change.

ELIGIBILITY:
Inclusion Criteria:

* Female
* First or second trimester of pregnancy
* First or second pregnancy
* Resident in the study area

Exclusion Criteria:

- Refuse to give informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2766 (Actual)
Dates: Start 2004-03; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Birth weight | At delivery

SECONDARY OUTCOMES:
Anemia | At 32 weeks gestation and at delivery
Peripheral and placental parasitaemia | At 32 weeks gestation (peripheral) and at delivery (both)
Gestational age | At first antenatal visit

CONTACTS AND LOCATIONS:
Overall Officials: Sheick Coulibaly Oumar Coulibaly, MD PhD, Study Director — Directeur de la Biologie Médicale du Laboratoire National de Santé Publique; Umberto D'Alessandro, MD, Study Chair — Institute of Tropical Medicine
Locations (1):
- District Sanitaire, Boromo, Burkina Faso